CLINICAL TRIAL: NCT03577847
Title: Rural CT Examination and Thrombolytic Treatment for Stroke: An Observational Study of Medical and Health Economic Effects
Brief Title: Rural CT Examination and Thrombolytic Treatment for Stroke
Acronym: RURALCT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Extrastiftelsen (Other)
Responsible Party: Sponsor
Other Study IDs: REK 2017/102
Record Dates: First submitted 2018-01-09; First posted 2018-07-05 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Stroke
Keywords: Stroke, Thrombolysis, Rural CT
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Intervention group: Stroke patients investigated with rural CT scanning at HSS, Ål. Patients living in the municipalities of Hol, Ål, Gol, Hemsedal and Nes.
  Interventions: Diagnostic Test: Rural CT scanning
- 2: Control-group: Stroke patients with similar transportation time to hospital, but no access to rural CT scanning. Patients living in the municipalities of Nore- and Uvdal, Vang, Øystre and Vestre Slidre, Lesja, Vågå, Lom, Dovre, Skjåk and Sel.

INTERVENTIONS:
Diagnostic Test: Rural CT scanning — Rural computer tomography for acute stroke
  Other Names: Thrombolysis
  Groups: 1

SUMMARY:
To counteract long term sequelae from stroke, ultrarapid diagnosis and treatment, high quality multidiciplinary in-hospital care and optimal long term rehabilitation is required. In this study, the investigators are moving the essential first diagnosis and treatment out into the community close to where the patient live, thus shortening the all important time from debut of symptoms to thrombolytic treatment improving the prognosis of stroke patients.

DETAILED DESCRIPTION:
Stroke is an acute, potentially mutilating disease. To counteract long term sequelae three factors are essential: Ultrarapid diagnosis and treatment, high quality multidiciplinary in-hospital care and optimal long term rehabilitation. Initial diagnosis and treatment has up to now been completed within the hospital domain. This study will change that: moving the essential first diagnosis and treatment out into the community close to where the patient lives thus shortening the all important time from debut of symptoms to thrombolytic treatment. We will operate a local computer tomography (CT) service in the hands of community based non-specialized health care personnel (MD and nurse) acting under direct telemetric guidance from on call hospital specialists. Thus, the investigators will show that by combining current technological advances in real time video communication with an acutely well functioning cooperation between the community and hospital health service personnel the prognosis of stroke patients is improved.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years being investigated by CT within 24 hours for acute symptoms of stroke.
2. Fullfilling criteria for the diagnosis acute stroke as described by the Norwegian stroke registry.
3. Giving informed consent.

Exclusion Criteria:

1. Symptoms not due to ischaemic or haemorrhagic stroke as adjudicated at discharge.
2. Not able to cooperate to 3 months follow up.
3. Not giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intervention group (access to local CT):
  Patients from the municipalities Hol, Ål, Gol, Hemsedal and Nes.
  Control group (no local CT):
  Patients from the municipalities Nore and Uvdal, Vang, Øystre- and Vestre Slidre, Lesja, Skjåk, Lom, Dovre, Vågå and Sel.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Thrombolytic treatment | 3 months
  The proportion of patients with ischaemic stroke receiving thrombolytic treatment in percent.

SECONDARY OUTCOMES:
Ictus to needle time | 3 months
  Time from onset of stroke symptoms (Ictus) to thrombolytic treatment (Needle).
Functional status | 3 months
  Modified Rankin Scale (mRS score 0-6). Good outcome 0-2
Cognitive status | 3 months
  Montreal Cognitive Assessment (MoCA score 0-30). Good outcome 26-30
Depression | 3 months
  Geriatric depression scale (GDS score 0-30). Good outcome 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Jorgen M Ibsen, MD, Principal Investigator — Vestre Viken Hospital Trust
Locations (1):
- Vestre Viken Hospital Trust, Hønefoss, Buskerud, Norway

IPD SHARING:
Plan to Share IPD: No